CLINICAL TRIAL: NCT06923241
Title: Nutri-score Labelling in a UK Restaurant Setting: a Randomised Control Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: University of Bristol (Other); Liverpool John Moores University (Other)
Responsible Party: Principal Investigator, Eric Robinson, Professor, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NS in the OOHFS study
Record Dates: First submitted 2025-03-26; First posted 2025-04-11 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: PME; Food Choice; Food Labelling
Keywords: Nutri-score; PME; Food choice

STUDY DESIGN:
Who Masked: Participant
Masking Description: To attempt to reduce the likelihood of aim guessing, participants will be recruited to a study described as 'A study of consumer behaviour in different restaurants'.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restaurant 1 (Active Comparator): Restaurant 1: plant-based cafe
  Interventions: Behavioral: menu labelling type
- Restaurant 2 (Active Comparator): Restaurant 2: University cafe
  Interventions: Behavioral: menu labelling type

INTERVENTIONS:
Behavioral: menu labelling type — Participants will be given a restaurant's menu with calorie information or a menu with calorie information and NS labelling.

SUMMARY:
An experiment exploring the perceived effectiveness of Nutri-score food labels with calorie labelling compared to calorie labelling only on food choice and consumption in a real-world setting

ELIGIBILITY:
Inclusion Criteria:

* Can visit a restaurant in Liverpool city centre
* Regularly eat food prepared out of the home (from restaurants, cafes, fast food etc., at least once a month)
* Over the age of 18 years
* Fluent English speaker

Exclusion Criteria:

* Pregnant/breastfeeding
* You have been diagnosed with a current or historic eating disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Perceived Message Effectiveness | Up to 30 weeks
  An adapted version of the University of North Carolina PME scale will be used to measure health concern, product attitude, and discouragement of item consumption in response to the food menu. Participants will be given the menu they ordered from to look at. All participants will answer 3 questions using a Likert scale ranging from 1 - 5 anchored by "not at all" and "a great deal". The mean response to the three items will be calculated. PME is used as an early indicator of a health message's potential to change behaviour (e.g., reduce selection of less healthy items). The scale has been used previously to identify the potential impact of food labels and is predictive of long-term behaviour.
Nutritional quality of each item and for the full meal | Up to 30 weeks
  Nutritional quality for meal choices will be calculated using the UK NPM scoring system. This calculates a score (continuous variable) for a product by deducting a total score for positive nutrients from a total score for negative nutrients. A lower score represents greater nutritional quality and a higher score represents poorer nutritional quality.
  We will calculate the mean NPM score weighted by energy content of items for each participant. This will ensure that the NPM score of main dishes will be weighted higher than that of starters or sides (assuming energy content of selected main is higher than any starters or sides), leading to a more representative overall NPM score for food orders. This will be done using the weighted.mean function in R. This function multiplies each value (i.e. NPM scores for individual items) by its corresponding weight (kcal content of individual items), sums all items and then divides this by the sum of the weights.

SECONDARY OUTCOMES:
NS label of each item selected | Up to 30 weeks
  A NS category value will be recorded for each item selected by participants (A,B,C,D,E)
Energy content of all food ordered | Up to 30 weeks
  The sum of energy (kcal) across all foods ordered for the meal will be calculated
Energy and nutrients consumed | Up to 30 weeks
  Researchers will take pictures of plates before and after each item is given to participants. Researchers will estimate the percentage of each dish consumed.
  Participants will be asked whether they shared any of their meal with someone else and this will be taken into account when making percentage estimates. A random 10% of percentage estimates will be performed by a second researcher to measure reliability.
  Energy and nutrient consumption will be calculated by multiplying the total energy/nutritional content of food items selected/consumed by the estimated proportion of the item consumed. Nutrients explored will be salt, sugar, fat, saturated fat, protein and fibre.
Later intake | Up to 30 weeks
  The morning after participants take part in the study, they will be emailed with a link to complete a dietary recall survey (via intake 24, https://intake24.co.uk/). Participants will report everything they ate after the study session up until they went to bed. They will be asked to provide as much detail as possible on what they had for dinner, snacks, and drinks after the study session. We will estimate based on data from Intake 24, later consumption (kcal, salt, fat, saturated fat, sugar, protein, fibre).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Robinson, Principal Investigator — University of Liverpool
Locations (1):
- University of Liverpool, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised participant data will be placed on the Open Science Framework in case other researchers want to use in the future.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD and supporting information will be available once the study is completed and published, with no end date.
Access Criteria: The IPD and supporting information will be uploaded to the Open Science Framework where it will be openly available.

DOCUMENTS (1):
  • Study Protocol (2025-04-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT06923241/Prot_000.pdf